CLINICAL TRIAL: NCT04184414
Title: CD19-CART Cells in the Treatment of CD19+ r/r B Cell-derived Hematological Malignancies
Brief Title: The Clinical Application of Chimeric Antigen Receptor T Cells in the Treatment of CD19 Positive Recurrent Refractory B Cell-derived Hematological Malignancies
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: PersonGen BioTherapeutics (Suzhou) Co., Ltd. (Industry)
Collaborators: Second Affiliated Hospital of Suzhou University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PA-P19-001
Record Dates: First submitted 2019-11-04; First posted 2019-12-03 (Actual); Last update posted 2019-12-03 (Actual); Status verified 2019-12

CONDITIONS: B Acute Lymphoblastic Leukemia; Mantle Cell Lymphoma; Follicular Lymphoma
MeSH Terms: conditions — Burkitt Lymphoma; Lymphoma, Mantle-Cell; Lymphoma, Follicular

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- CART cells (Experimental): dosage：Once dose，1.0*10^6cells/kg CART cells Administration mode:Intravenous infusion
  Interventions: Drug: CD19-CART

INTERVENTIONS:
Drug: CD19-CART — 1-10x106 / kg CD19 CART cells
  Other Names: Targeting hcd19 chimeric antigen receptor

SUMMARY:
CD19 is expressed in most B malignant tumors, especially in the former B cells ALL. This makes CD19 a natural target of immunotherapy. In terms of safety, the lack of B cells caused by CD19 targeted therapy will not cause life-threatening side effects (of course, Ig supplementation is necessary in the long-term B cell inhibition therapy). Moreover, the number of B cells can be restored after removing anti-CD19 treatment measures (such as anti-CD19 CART cells). In addition, CD19 has been chosen as the target of B-ALL therapy for the following reasons: ① as the BCR signal "amplifier", CD19 plays a role in PAX-5-mediated tumor formation; ② by activating MYC (as the oncogene controlled by PAX-5, C-MYC plays a key role in promoting the malignant proliferation of B cells), CD19 can cause B-ALL formation. Based on the above reasons, CD19 has become an ideal target in the treatment of B-cell cancer.

ELIGIBILITY:
Inclusion Criteria:

* 1. At the time of initial diagnosis, the age is 18-70 years old, regardless of gender or race
* 2. Morphological analysis showed that the load of lymphoma was ≥ 5%
* 3. Estimated survival time > 12 weeks
* 4. The main investigator and the attending physician of the patient think that there is no other feasible and effective alternative treatment, such as hematopoietic stem cell transplantation
* 5. Relapsed / refractory B-cell acute lymphocytic leukemia (all): A. objective remission rate (or) of grade 2 or higher bone marrow recurrence B. bone marrow relapse after allogeneic stem cell transplantation (SCT), SCT treatment is more than 6 months and in or state before cart-19 reinfusion C. refractory patients (CR status is not reached after 2 rounds of standard chemotherapy (CR refers to the load of myeloma detected by morphology < 5%)) D. Philadelphia chromosome positive (Ph +) and tyrosine kinase inhibitor (TKI) treatment failed twice or TKI failed to maintain or E. treatment with allogeneic SCT
* 6. For patients with relapse, CD19 was detected in bone marrow or peripheral blood by flow cytometry within 3 months before admission
* 7. CD19 expression on lymphoma cells: immunohistochemistry > 15% or flow cytometry > 30%
* 8. The main organ functions are sound, including: A. renal function: radioisotope glomerular filtration rate > 60 ml / min / 1.73 m2, or serum creatinine clearance rate in line with relevant age / gender standards B. alanine transferase (ALT) < 5 times the normal maximum value of the same age C. bilirubin < 2.0 mg / dl D. to achieve the minimum pulmonary function: ≤ grade I dyspnea and indoor blood oxygen concentration > 91% E. echocardiography or multi gated angiography (MUGA) showed that the left ventricular short axis shortening rate (LVSF) was ≥ 28%, or left ventricular ejection fraction (LVEF) was ≥ 45%
* 9. Karnofsky score (age ≥ 16 years old) ≥ 50 or zubrod-ecog-who score ≤ 2
* 10. Sign written informed consent and obtain consent before any research is carried out
* 11. When the above other conditions are met, the cell culture factory must receive fresh blood samples from patients. In the case of monocultured cells, they can only be accepted by the cell culture factory if the relevant tests are qualified

Exclusion Criteria:

* 1. Recurrence of isolated extramedullary diseases
* 2. The patient is accompanied by the following genetic syndrome: Fanconi syndrome, Kostmann syndrome, Shwachman syndrome or any known myelofailure syndrome. Patients with Down syndrome are not included in the exclusion criteria
* 3. Patients with Burkitt's lymphoma / leukemia (i.e. patients with mature B cell all, B cell surface immunoglobulin positive (SIG +) and light chain kappa or lambda type, morphology Fab L3 or myc ectopic expression)
* 4. Patients with previous history of malignant tumor but cured skin or cervical carcinoma in situ and patients with inactive tumor are not included in the exclusion criteria
* 5. Previous use of gene therapy
* 6. Previous use of anti-CD19 / CD3 combination therapy or any other anti-CD19 treatment
* 7. Hepatitis B or C or HBV / HCV or other uncontrolled infection at the time of screening
* 8. Screening with HIV infection
* 9. Acute or chronic graft-versus-host reaction (GVHD) of level 2-4
* 10. Use the following drugs: A. steroid: it is forbidden to use within 72 hours before cart-19 reinfusion, but physiological steroid treatment dose (< 6 - 12 mg / m2 / day) or equivalent hydrocortisone can be used B. allogeneic cell therapy: no donor lymphocyte infusion (DLI) is allowed within 6 weeks before cart-19 reinfusion C. GVHD treatment: any GVHD treatment (such as calmodulinase inhibitor, methotrexate, mycophenolate ester, steroid (see above), rapamycin, thalidomide or immunosuppressive antibody (such as anti-CD20 / TNF / IL6 / IL6R)) must be stopped within 4 weeks before cart-19 infusion D. chemotherapy: I. The following drugs should be stopped for at least one week before cart-19 infusion, and it is better not to accompany or follow the lymphocyte elimination chemotherapy plan: hydroxyurea, vincristine, 6-mercaptopurine, 6-thioguanine, methotrexate < 25 mg / m2, cytarabine < 10 mg / m2 / day, asparaginase; II. The following drugs should be stopped for at least four weeks before cart-19 infusion: remedial chemotherapy (such as chlorine method) Lapin, cytarabine > 100 mg / m2, anthracycline drugs, cyclophosphamide), lymphocyte clearance chemotherapy drugs are not included in the exclusion criteria E. central nervous system (CNS) disease prevention: CNS prevention and treatment should be stopped at least one week before cart-19 reinfusion (such as MTX injection into spinal cord)
* 11. For CNS infiltration of malignant tumors, refer to the guidelines of national comprehensive cancer network (NCCN) cns-3. Note: the patients with CNS diseases who have been effectively treated are not included in the exclusion criteria. The patients cannot participate in the drug trial within 30 days before screening
* 12. Pregnant or lactating women: 48 hours before reinfusion, the female test participants must carry out serum or urine pregnancy test, and the test result is positive
* 13. Women of childbearing age and all men did not take effective contraceptive methods within one year after cart-19 transfusion

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2018-01-09 (Actual); Primary Completion 2020-01-01 (Estimated); Study Completion 2020-01-01 (Estimated)

PRIMARY OUTCOMES:
CR | 12 weeks after infusion of the study drug
  Complete response rate (CR)

SECONDARY OUTCOMES:
PR | 12 weeks after infusion of the study drug
  Partial remission rate
2-year disease-free survival rate 2-year disease-free survival rate | 12 weeks after infusion of the study drug
  2-year disease-free survival rate

CONTACTS AND LOCATIONS:
Locations (1):
- Hematology Department of the Second Affiliated Hospital of Suzhou University, Suzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No